CLINICAL TRIAL: NCT02410278
Title: A Multicenter, Double- Blind, Placebo- Controlled Study of Montelukast on Gastrointestinal Tolerability in Patients With Relapsing Forms of Multiple Sclerosis Receiving Tecfidera® (Dimethyl Fumarate) Delayed Release Capsules
Brief Title: Study of Montelukast on Gastrointestinal Tolerability in Patients With Relapsing Forms of Multiple Sclerosis Receiving Tecfidera
Acronym: MITIGATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 109MS414
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMF plus montelukast (Experimental): DMF as described in the United States Prescribing Information (USPI) plus 10mg montelukast tablet once daily according to the prevailing product label (Singulair)
  Interventions: Drug: dimethyl fumarate; Drug: montelukast
- DMF plus placebo (Experimental): DMF as described in the USPI plus matched placebo
  Interventions: Drug: dimethyl fumarate; Drug: Placebo

INTERVENTIONS:
Drug: dimethyl fumarate — Starting dose of 120 mg twice daily orally After 7 days, maintenance dose of 240 mg twice daily orally
  Other Names: BG00012; Tecfidera; DMF
Drug: montelukast — As described in the treatment arm
  Other Names: Singulair
  Arms: DMF plus montelukast
Drug: Placebo — Matched placebo
  Arms: DMF plus placebo

SUMMARY:
The primary objective of this study is to evaluate whether montelukast can reduce the severity of gastrointestinal (GI) events, measured by the Gastrointestinal Symptom Rating Scale (GSRS), after oral administration of dimethyl fumarate (DMF) in participants with relapsing forms of Multiple Sclerosis (MS). The secondary objectives of this study are as follows: To evaluate whether montelukast after oral administration of DMF in participants with relapsing forms of MS decreases discontinuations due to GI events and reduces the number of participants taking symptomatic therapies for GI events; To investigate the effect of montelukast on the incidence of flushing events after oral administration of 240 mg DMF in participants with relapsing forms of MS.

ELIGIBILITY:
Key Inclusion Criteria:

* Reside in the United States and have a confirmed diagnosis of a relapsing form of MS and satisfy the therapeutic indication as described in the local label
* As perceived by the Investigator, have the ability to comply with all requirements of the study protocol and to operate the eDiary required to record GI-related events
* Female participants of childbearing potential who are not surgically sterile must practice effective contraception during their participation in the study and be willing and able to continue contraception for 30 days after they complete or withdraw from the study. All men must practice effective contraception, and they should not donate sperm throughout the study and for at least 90 days after their last dose of study treatment.

Key Exclusion Criteria:

* History of significant GI disease (for example, irritable bowel disease, peptic ulcer disease, history of major GI surgery, eosinophilic GI disease, or food allergies)
* Chronic use (≥7 consecutive days) of bismuth subsalicylate, simethicone, calcium carbonate, loperamide, proton-pump inhibitors, or ondansetron within 1 month prior to the Screening Visit
* Use of the following medications: montelukast, immunotherapy, mast cell stabilizers, or parenteral, inhaled, or oral steroids up to 1 month prior to the Screening Visit. Use of these medications is also not permitted for the duration of the study (except for the use of montelukast as per study protocol) and will lead to discontinuation
* Have one or more major comorbidities that, in the opinion of the Investigator, may affect the outcome of the study
* History of malignancy (except for basal cell carcinoma that had been completely excised prior to study entry), severe allergic or anaphylactic reactions or known drug hypersensitivity, abnormal laboratory results indicative of any significant disease, and/or a major disease that would preclude participation in a clinical study

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (49):
- United States (49):
  - Research Site, Jonesboro, Arkansas
  - Research Site, Carmichael, California
  - Research Site, La Jolla, California
  - Research Site, La Mesa, California
  - Research Site, Pomona, California
  - Research Site, Simi Valley, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fairfield, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Naples, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Rome, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Flossmoor, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Scarborough, Maine
  - Research Site, Farmington Hills, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Freehold, New Jersey
  - Research Site, Amherst, New York
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, Hendersonville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Sanford, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Tualatin, Oregon
  - Research Site, Dickson City, Pennsylvania
  - Research Site, Greensburg, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Wilkes-Barre, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Alexandria, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 50 sites in the United States.
Pre-assignment Details: Participants were screened over 2 weeks. Those who met ≥1 of the following criteria were considered screen failures: a score of ≥5 on 1 question for 1 day on the Gastrointestinal Symptom Rating Scale (GSRS), ≥4 or ≥3 on 1 question for 2 or 3 consecutive days, respectively; and eDiary compliance of <75% over 14 days prior to randomization.
Groups:
- Dimethyl Fumarate (DMF)- Run-in Period: Participants received 120 milligrams (mg) of DMF twice daily by mouth for 7 days and 240 mg twice daily (as described in the USPI) for up to 28 days. Participants who reached the predefined threshold in scores on the GSRS continued to the Study Treatment Period; all other participants were discontinued from the study.
- Placebo- Study Treatment: Participants who reached the predefined threshold in scores on the GSRS during the Run-in Period entered the Study Treatment Period. Participants continued to receive 240 mg DMF twice daily and also received a montelukast-matching placebo tablet once daily by mouth for 8 weeks. Participants received only 240 mg DMF twice daily for 2 weeks after discontinuing treatment with placebo, then were followed for 2 additional weeks before a final phone interview.
- Montelukast- Study Treatment: Participants who reached the predefined threshold in scores on the GSRS during the Run-in Period entered the Study Treatment Period. Participants continued to receive 240 mg DMF twice daily and also received 10 mg of montelukast once daily by mouth for 8 weeks. Participants received only 240 mg DMF twice daily for 2 weeks after discontinuing treatment with montelukast, then were followed for 2 additional weeks before a final phone interview.
Period: Run-in Period
Arm/Group | Dimethyl Fumarate (DMF)- Run-in Period | Placebo- Study Treatment | Montelukast- Study Treatment
Started | 102 | 0 | 0
Received at Least 1 Dose of DMF | 98 | 0 | 0
Completed | 64 | 0 | 0
Not Completed | 38 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — GSRS Threshold Not Met | 30 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Period: Study Treatment Period
Arm/Group | Dimethyl Fumarate (DMF)- Run-in Period | Placebo- Study Treatment | Montelukast- Study Treatment
Started | 0 | 31 | 33
Modified Intent-to Treat(mITT)Population | 0 | 30 | 33
Completed Randomized Study Treatment | 0 | 20 | 29
Completed | 0 | 20 | 29
Not Completed | 0 | 11 | 4
Not completed — Adverse Event | 0 | 6 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Other | 0 | 3 | 0
Not completed — GSRS Threshold Not Met | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The MITT: All participants who were randomized, received at least 1 dose of DMF treatment, received at least 1 dose of study treatment (montelukast or placebo) on/after the first DMF dose date, and had at least 1 GSRS score measurement during the Day 1 - Day 10 period.
Groups:
- MITT- Placebo: Participants who reached the predefined threshold in scores on the GSRS during the Run-in Period entered the Study Treatment Period. Participants continued to receive 240 mg DMF twice daily and also received a montelukast-matching placebo tablet once daily by mouth for 8 weeks. Participants received only 240 mg DMF twice daily for 2 weeks after discontinuing treatment with placebo, then were followed for 2 additional weeks before a final phone interview. One participant randomized to placebo was excluded from the MITT.
- MITT-Montelukast: Participants who reached the predefined threshold in scores on the GSRS during the Run-in Period entered the Study Treatment Period. Participants continued to receive 240 mg DMF twice daily and also received 10 mg of montelukast once daily by mouth for 8 weeks. Participants received only 240 mg DMF twice daily for 2 weeks after discontinuing treatment with montelukast, then were followed for 2 additional weeks before a final phone interview.
- Total: Total of all reporting groups
Arm/Group | MITT- Placebo | MITT-Montelukast | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.63 (13.00) | 44.88 (10.39) | 44.29 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Worsening in Severity of Gastrointestinal (GI) Adverse Events (AEs) on the GSRS From Day 0 to Day 10
Description: The GSRS is a weekly recall scale that was modified for daily recall. The 15-question GSRS is summarized with a 7-point Likert scale: no discomfort at all=0; minor discomfort=1; mild discomfort=2; moderate discomfort=3; moderately severe discomfort=4; severe discomfort=5 and very severe discomfort=6. The overall GSRS score is a mean score that ranges from 0 (no symptoms) to 6 (the worst possible symptoms). Worsening in severity was defined as a positive average change from baseline (Day 0) to Day 10 in the GSRS score. Day 0: the day before a participant started randomized treatment (if the GI threshold was reached 1 day previously) or the first day of randomized treatment if the threshold was reached that day. If the threshold was reached >1 day previously, then Day 0 was the last day when the threshold was reached, prior to the first dose. Average change is the sum of changes from baseline in GSRS score over the first 10 days divided by the total of days with a GSRS score.
Time Frame: Baseline (Day 0), Day 10 (10 days after Day 0)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- MITT-Placebo: Participants who reached the predefined threshold in scores on the GSRS during the Run-in Period entered the Study Treatment Period. Participants continued to receive 240 mg DMF twice daily and also received a montelukast-matching placebo tablet once daily by mouth for 8 weeks. Participants received only 240 mg DMF twice daily for 2 weeks after discontinuing treatment with placebo, then were followed for 2 additional weeks before a final phone interview. One participant randomized to placebo was excluded from the MITT.
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
percentage of participants | 17 | 33
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Odds ratio is the odds of an event in the Montelukast treatment group divided by the odds of an event in the placebo treatment group. P-value is from the likelihood ratio test that the odds ratio is 1. CI = profile likelihood confidence interval; Test type: Superiority; p = 0.0617, weighted logistic regression model; Odds Ratio (OR) = 3.931, 95% CI 2-sided [0.938 to 20.832]

2. Secondary Outcome: Average Change From Baseline in GSRS Overall Score at Day 1 to Day 10
Description: The GSRS is a weekly recall scale that was modified for daily recall. The 15-question GSRS is summarized with a 7-point Likert scale: no discomfort at all=0; minor discomfort=1; mild discomfort=2; moderate discomfort=3; moderately severe discomfort=4; severe discomfort=5 and very severe discomfort=6. The overall GSRS score is a mean score that ranges from 0 (no symptoms) to 6 (the worst possible symptoms). This endpoint reports the average change from baseline (Day 0) at Day 1 to Day 10. Day 0: the day before a participant started randomized treatment (if the GI threshold was reached 1 day previously) or the first day of randomized treatment if the threshold was reached that day. If the threshold was reached >1 day previously, then Day 0 was the last day when the threshold was reached, prior to the first dose. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline (Day 0), Day 1 (1 day after Day 0), Day 10 (10 days after Day 0)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
units on a scale
  Day 0 | 0.80 (0.569) | 0.84 (0.576)
  Change From Day 1 to Day 10 | -0.28 (0.695) | -0.23 (0.499)
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Results are obtained from an ANCOVA model for comparing average change of the GSRS score in the two treatment groups, adjusted for age, weight and baseline GSRS score. Weights, defined as the proportions of days with GSRS score recorded during the Day 1 - Day 10 period are applied to adjust for missing data; Test type: Superiority; p = 0.3753, ANCOVA; adjusted mean difference = 0.084, 95% CI 2-sided [-0.104 to 0.273]

3. Secondary Outcome: Average Change From Baseline in GSRS Overall Score at Day 1 to Week 10
Description: The GSRS is a weekly recall scale that was modified for daily recall. The 15-question GSRS is summarized with a 7-point Likert scale: no discomfort at all=0; minor discomfort=1; mild discomfort=2; moderate discomfort=3; moderately severe discomfort=4; severe discomfort=5 and very severe discomfort=6. The overall GSRS score is a mean score that ranges from 0 (no symptoms) to 6 (the worst possible symptoms). This endpoint reports the average change from baseline (Day 0) between Day 1 and Week 10. Day 0: the day before a participant started randomized treatment (if the GI threshold was reached 1 day previously) or the first day of randomized treatment if the threshold was reached that day. If the threshold was reached >1 day previously, then Day 0 was the last day when the threshold was reached, prior to the first dose. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline (Day 0), Day 1 (1 day after Day 0), Week 10 (10 weeks after Day 0)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
units on scale
  Day 0 | 0.80 (0.569) | 0.84 (0.576)
  Change From Day 1 to Week 10 | -0.37 (0.67) | -0.31 (0.55)
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and Week 10; Test type: Superiority; p = 0.0376, Repeated measures model; adjusted mean difference = 0.081, 95% CI 2-sided [0.005 to 0.158]

4. Secondary Outcome: Time to First Worsening From Baseline in GSRS Overall Score at Day 1 to Day 10
Description: The GSRS is a weekly recall scale that was modified for daily recall. The 15-question GSRS is summarized with a 7-point Likert scale: no discomfort at all=0; minor discomfort=1; mild discomfort=2; moderate discomfort=3; moderately severe discomfort=4; severe discomfort=5 and very severe discomfort=6. The overall GSRS score is a mean score that ranges from 0 (no symptoms) to 6 (the worst possible symptoms). Day 0: the day before a participant started randomized treatment (if the GI threshold was reached 1 day previously) or the first day of randomized treatment if the threshold was reached that day. If the threshold was reached >1 day previously, then Day 0 was the last day when the threshold was reached, prior to the first dose.. Time to the first worsening was defined as the number of days from Day 1 to the first date with a worsened GSRS score. Censoring occurred at Day 10.
Time Frame: Baseline (Day 0), Day 1 (1 day after Day 0) to Day 10 (10 days after Day 0)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
days | 10 [3 to NA] — The upper limit of the inter-quartile range was not estimated because the Kaplan Meier curve did not cross the 75th percentile threshold during the 10 days of data collection for this outcome measure. | 7 [1 to NA] — The upper limit of the inter-quartile range was not estimated because the Kaplan Meier curve did not cross the 75th percentile threshold during the 10 days of data collection for this outcome measure.
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Hazard ratio and the P-value are based on the Cox's proportional hazard regression model, adjusted for age, weight and baseline GSRS score. Hazard ratio (HR) is the ratio of hazard rates of Montelukast and placebo treatment groups. P-value is from the Wald test that HR is 1. CI = Wald confidence interval; Test type: Superiority; p = 0.7952, Regression, Cox; Hazard Ratio (HR) = 1.094, 95% CI 2-sided [0.554 to 2.164]

5. Secondary Outcome: Time to Recovery to Baseline GSRS Score From Last Occurrence of Worst GSRS Score at Day 1 to Week 8
Description: The GSRS is a weekly recall scale that was modified for daily recall. The 15-question GSRS is summarized with a 7-point Likert scale: no discomfort at all=0; minor discomfort=1; mild discomfort=2; moderate discomfort=3; moderately severe discomfort=4; severe discomfort=5 and very severe discomfort=6. The overall GSRS score is a mean score that ranges from 0 (no symptoms) to 6 (the worst possible symptoms). Recovery was defined as a GSRS score less than or equal to the Day 0 score. Day 0: the day before a participant started randomized treatment (if the GI threshold was reached 1 day previously) or the first day of randomized treatment if the threshold was reached that day. If the threshold was reached >1 day previously, then Day 0 was the last day when the threshold was reached, prior to the first dose. Time to recovery was defined as the date of recovery minus the date of the last occurrence of the worst score.
Time Frame: Baseline (Day 0), Day 1 (1 Day after Day 0) to Week 8 (8 weeks after Day 0)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
days | 1 [1 to 3] | 1 [1 to 2]
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.8328, Regression, Cox; Hazard Ratio (HR) = 0.946, 95% CI 2-sided [0.563 to 1.589]

6. Secondary Outcome: Average Change From Baseline in GSRS Overall Score at Day 1 to Weeks 1 to 8
Description: The GSRS is a weekly recall scale that was modified for daily recall. The 15-question GSRS is summarized with a 7-point Likert scale: no discomfort at all=0; minor discomfort=1; mild discomfort=2; moderate discomfort=3; moderately severe discomfort=4; severe discomfort=5 and very severe discomfort=6. The overall GSRS score is a mean score that ranges from 0 (no symptoms) to 6 (the worst possible symptoms). This endpoint reports the average change from baseline (Day 0) between Day 1 and the specified time point. Day 0: the day before a participant started randomized treatment (if the GI threshold was reached 1 day previously) or the first day of randomized treatment if the threshold was reached that day. If the threshold was reached >1 day previously, then Day 0 was the last day when the threshold was reached, prior to the first dose. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline (Day 0), Day 1 (1 Day after Day 0), Weeks 1 to 8 (1-8 weeks after Day 0)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
unit on scale
  Day 0 | 0.80 (0.569) | 0.84 (0.576)
  Change from Day 1 to Week 1 | -0.30 (0.686) | -0.21 (0.498)
  Change from Day 1 to Week 2 | -0.29 (0.701) | -0.25 (0.495)
  Change from Day 1 to Week 3 | -0.31 (0.686) | -0.26 (0.522)
  Change from Day 1 to Week 4 | -0.33 (0.679) | -0.26 (0.537)
  Change from Day 1 to Week 5 | -0.35 (0.674) | -0.28 (0.533)
  Change from Day 1 to Week 6 | -0.35 (0.673) | -0.29 (0.537)
  Change from Day 1 to Week 7 | -0.36 (0.673) | -0.30 (0.544)
  Change from Day 1 to Week 8 | -0.36 (0.677) | -0.31 (0.548)
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 1: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.1743, Repeated measures model; adjusted mean difference = 0.115, 95% CI 2-sided [-0.052 to 0.283]
Statistical Analysis 2: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 2: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.2677, Repeated measures model; adjusted mean difference = 0.079, 95% CI 2-sided [-0.063 to 0.221]
Statistical Analysis 3: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 3: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.1788, Repeated measures model; adjusted mean difference = 0.085, 95% CI 2-sided [-0.040 to 0.211]
Statistical Analysis 4: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 4: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.0866, Repeated measures model; adjusted mean difference = 0.100, 95% CI 2-sided [-0.015 to 0.216]
Statistical Analysis 5: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 5: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.0509, Repeated measures model; adjusted mean difference = 0.100, 95% CI 2-sided [-0.000 to 0.201]
Statistical Analysis 6: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 6: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.0649, Repeated measures model; adjusted mean difference = 0.088, 95% CI 2-sided [-0.006 to 0.182]
Statistical Analysis 7: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 7: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.0479, Repeated measures model; adjusted mean difference = 0.088, 95% CI 2-sided [0.001 to 0.176]
Statistical Analysis 8: Comparison: MITT-Placebo vs MITT-Montelukast; Change from Day 1 to Week 8: Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight(kg) and baseline GSRS score, and has spatial-exponential variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and the specified time point; Test type: Superiority; p = 0.0540, Repeated measures model; adjusted mean difference = 0.082, 95% CI 2-sided [-0.001 to 0.166]

7. Secondary Outcome: Average Change From Baseline in GSRS Overall Score at Day 0 to 72 Hours From the Initiation of Randomized Study Treatment
Description: The GSRS is a weekly recall scale that was modified for daily recall. The 15-question GSRS is summarized with a 7-point Likert scale: no discomfort at all=0; minor discomfort=1; mild discomfort=2; moderate discomfort=3; moderately severe discomfort=4; severe discomfort=5 and very severe discomfort=6. The overall GSRS score is a mean score that ranges from 0 (no symptoms) to 6 (the worst possible symptoms). This endpoint reports the average change from baseline (Day 0) at Day 1 to Day 3. Day 0: the day before a participant started randomized treatment (if the GI threshold was reached 1 day previously) or the first day of randomized treatment if the threshold was reached that day. If the threshold was reached >1 day previously, then Day 0 is the last day when the threshold was reached, prior to the first dose. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline (Day 0), Day 3 (72 hours after Day 0)
Population: The MITT: All participants who were randomized, received at least 1 dose of both DMF treatment and study treatment (montelukast or placebo) on/after the first DMF dose date, and had at least 1 GSRS score measurement during the Day 1 - Day 10 period. One participant in the MITT-Montelukast arm did not provide post-baseline data.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
units on scale
  Day 0 | 0.80 (0.569) | 0.84 (0.576)
  Change from Day 0 to Day 3: number analyzed (Participants) | 30 | 32
  Change from Day 0 to Day 3 | -0.28 (0.665) | -0.18 (0.528)
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Results are obtained from a repeated measures model for change from baseline (Day 0) in the GSRS score. The model includes treatment, day and treatment by day interaction, adjusted for age, weight (kg) and baseline GSRS score, and has unstructured variance-covariance structure. The P-value is for testing the null hypothesis of no difference between the two treatment groups in the average change from baseline (Day 0) between Day 1 and Day 3; Test type: Superiority; p = 0.2469, Repeated measures model; adjusted mean difference = 0.129, 95% CI 2-sided [-0.092 to 0.349]

8. Secondary Outcome: Percentage of Participants Who Required GI Symptomatic Therapy During the Study
Description: Symptomatic therapies were not permitted during the first 10 days after starting montelukast or placebo. From Day 10 onward, participants were allowed to use the following symptomatic therapies to treat DMF-related GI events: bismuth subsalicylate, simethicone, calcium carbonate, loperamide, proton-pump inhibitors and ondansetron.
Time Frame: Day 10 to Week 10
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
percentage of participants | 33 | 33
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Test type: Superiority; p = 1.0000, Chi-squared

9. Secondary Outcome: Percentage of Participants Who Discontinued DMF Therapy Due to GI-Related Adverse Events (AEs) From Day 0 to Week 10
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. Participants used an electronic diary to record GI-related events. GI-related AEs included diarrhea, nausea, upper abdominal pain, abdominal pain, and dyspepsia.
Time Frame: Day 0 to Week 10
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
percentage of participants | 7 | 9
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Test type: Superiority; p = 1.0000, Fisher's Exact

10. Secondary Outcome: Percentage of Participants Who Experienced AEs Related to Flushing
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. Flushing-related AEs included flushing and hot flush. Only events with an onset date on or after the date of first DMF dose (up to 27 days before Day 0) are presented. This includes events present before and subsequently worsened after the first dose of DMF.
Time Frame: Day of first DMF dose (up to 27 days before Day 0) to Week 10
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | MITT-Placebo | MITT-Montelukast
Number analyzed (Participants) | 30 | 33
percentage of participants | 23 | 36
Statistical Analysis 1: Comparison: MITT-Placebo vs MITT-Montelukast; Test type: Superiority; p = 0.2604, Chi-squared

ADVERSE EVENTS:
Time Frame: AEs were assessed for up to 16 weeks for the DMF Safety Population and for 8 weeks for the Primary Safety Population.
Groups:
- DMF Safety Population: Participants who received at least 1 dose of DMF.
- Primary Safety Population-Placebo: Participants who received at least 1 dose of placebo during the Study Treatment Period.
- Primary Safety Population-Montelukast: Participants who received at least 1 dose of montelukast during the Study Treatment Period.
Arm/Group | DMF Safety Population | Primary Safety Population-Placebo | Primary Safety Population-Montelukast
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 3/98 | 2/31 | 1/33
Other Adverse Events (participants affected / at risk) | 35/98 | 14/31 | 14/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DMF Safety Population (N=98) | Primary Safety Population-Placebo (N=31) | Primary Safety Population-Montelukast (N=33)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DMF Safety Population (N=98) | Primary Safety Population-Placebo (N=31) | Primary Safety Population-Montelukast (N=33)
Viral upper respiratory tract infection (Infections and infestations) | 10 | 5 | 4
Paraesthesia (Nervous system disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 5 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Liver function test increased (Investigations) | 0 | 0 | 2
Flushing (Vascular disorders) | 21 | 4 | 5
Fatigue (General disorders) | 5 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT02410278/Prot_SAP_000.pdf